CLINICAL TRIAL: NCT00108043
Title: Orthostatic Tolerance During FES-evoked Stepping in Paraplegia: A Safety and Viability Study
Brief Title: Orthostatic Tolerance During FES (Functional Electrical Stimulation)-Walking in Paraplegia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sydney (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHMRC 302013
Record Dates: First submitted 2005-04-12; First posted 2005-04-13 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Spinal Cord Injury
Keywords: Functional Electrical Stimulation; Gait; Blood pressure; Orthostatic Hypotension; Cardiovascular responses; Near-infra red spectroscopy
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic

INTERVENTIONS:
Procedure: FES-evoked functional upright gait

SUMMARY:
Objective:

The objective of this research is to undertake a safety and viability study of FES-evoked stepping in individuals with paraplegia. The rationale for this objective is based upon the need to clarify whether physiological limitations, especially orthostatic intolerance, limit functional mobility outcomes. The cardiovascular, autonomic, and muscle metabolic factors governing orthostatic tolerance during skin-surface FES stepping will be investigated, since this functional task forms the basis of upright mobility and engenders strong physiological challenges upon key regulatory processes in the SCI (spinal cord injury) patient.

Specific Hypotheses:

i. Reduction of blood pressure will be greater during FES-evoked stepping than during passive stepping; ii. Reduction of blood pressure will be greater during FES-evoked stepping with no upper body component versus FES-stepping with an upper body component; iii. Blood pressure will be reduced even further during FES-evoked stepping following a 6-week progressive-intensity gait training intervention.

DETAILED DESCRIPTION:
Aims:

The primary aim of the safety and viability study is to assess changes in blood pressure during up to 60-min of FES-evoked stepping versus up to 60-min of stepping.

A secondary aim is to investigate changes in blood pressure during FES-assisted stepping with and without a voluntary upper-limb component of gait.

Specific Hypotheses:

i. Reduction of blood pressure will be greater during FES-evoked stepping than during passive stepping; ii. Reduction of blood pressure will be greater during FES-evoked stepping with no upper body component versus FES-stepping with an upper body component; iii. Blood pressure will be reduced even further during FES-evoked stepping following a 6-week progressive-intensity gait training intervention.

Primary Outcome: The primary outcome measure for this study is the change of systolic blood pressure during three FES-evoked stepping conditions, as described below. Each condition is defined as up to 60-min of continuous gait.

Secondary Outcomes: Secondary outcomes include a change of diastolic blood pressure and the duration of orthostatic tolerance. Orthostatic tolerance will be assessed as the time that the subject can perform stepping before the onset of orthostatic hypotension. The duration of orthostatic tolerance will be determined by the time at which one of the following occur: (i) 60 continuous minutes of stepping; or (ii) orthostatic hypotension, defined as a reduction in systolic blood pressure of > 20 mmHg or diastolic blood pressure of >10 mmHg; or (iii) signs and symptoms of pre-syncope; or (iii) upon subject request. Throughout each trial, heart rate and blood pressure will be monitored continuously. In addition to the primary and secondary outcome variables, several additional measurements that may contribute to orthostatic tolerance, or indeed, intolerance, will be assessed at 10-min intervals during stepping.

ELIGIBILITY:
Inclusion Criteria:

* Male
* A spinal cord lesion, of traumatic etiology, between the 6th and 11th thoracic spinal segments
* Sensory and motor complete lesion (ASIA [American Spinal Injury Association]-A)
* At least 2 years post injury
* Between 18-55 years of age
* Responsive to electrical stimulation

Exclusion Criteria:

* Severe osteoporosis, fractures, dislocations (as determined by X-ray and DEXA)
* Upper limb or shoulder pathologies
* Severe spasticity (≥4 on Ashworth scale)
* Contractures
* Currently undertaking FES or gait training

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2004-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change of systolic blood pressure during three FES-evoked stepping conditions

SECONDARY OUTCOMES:
Cardiovascular and Metabolic Responses
Autonomic Responses
Muscle Metabolic Responses
Humoral Responses
Syncope Symptom Score

CONTACTS AND LOCATIONS:
Overall Officials: Glen M Davis, PhD, FACSM, Principal Investigator — University of Sydney
Locations (1):
- Rehabilitation Research Centre, University of Sydney, Sydney, New South Wales, Australia